CLINICAL TRIAL: NCT05247502
Title: Impact of the Characteristics of Acute Renal Failure in Intensive Care on the Long-term Renal Prognosis: Prospective Multicenter Cohort Study
Acronym: MAKI
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2021 LAUTRETTE; 2021-A01472-39 (Other: 2021-A01472-39)
Record Dates: First submitted 2022-02-09; First posted 2022-02-21 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Acute Kidney Injury; Transient Acute Renal Failure; Persistent Acute Renal Failure
Keywords: follow-up; intensive care unit; chronic kidney disease
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ICU patients without Acute Kidney Injury: Intensive care unit (ICU) patients who do not develop acute kidney injury (AKI) during their stay.
  AKI will be defined by KDIGO stage 1.
  The baseline serum creatinine (sCr) measurement will be defined as the sCr at admission if the corresponding estimation of glomerular filtration rate (GFR) by CKD-EPI formula is at least 90ml/min/1.73m2. Otherwise, the most recent sCr measured from 7-365 days prior to admission will be used. If there is no sCr measurement available from this period, it will be estimated using a reverse CKD-EPI formula for a GFR of 75 ml/min/1.73m2.
  No intervention is foreseen out of the observation of data relative to kidney function during ICU stay, at 3 month and 12 month of ICU admission.
  There will be no biological sample collection.
  Interventions: Biological: Data observation
- ICU patients with transient Acute kidney injury: Transient AKI will be defined as a complete renal recovery within 48 hours after the start of AKI.
  Complete renal recovery will be defined as a return to within 25% of the baseline serum creatinine measurement. TIf several AKI episodes occur during the patient's ICU stay, only the longest episode will be considered.
  No intervention is foreseen out of the observation of data relative to kidney function during ICU stay, at 3 month and 12 month of AKI start.
  There will be no biological sample collection.
  Interventions: Biological: Data observation
- ICU patients with persistent Acute kidney injury: If the AKI episode lasts longer than 48 hours, it will be classified as persistent AKI. If several AKI episodes occur during the patient's ICU stay, only the longest episode will be considered.
  No intervention is foreseen out of the observation of data relative to kidney function during ICU stay, at 3 month and 12 month of AKI start.
  There will be no biological sample collection.
  Interventions: Biological: Data observation

INTERVENTIONS:
Biological: Data observation — At the time of participant inclusion in the study, demographic data and a baseline serum creatinine measurement will be collected. During the patient's ICU stay, the occurrence and duration of any AKI episode will be recorded. Data related to diagnostic examinations of these AKI episodes will also be collected in accordance with practices guidelines. Data related to AKI monitoring will also be collected, including serum creatinine and urea daily follow-up measurements, diuresis, and nephrotoxic use. The patient's need for extrarenal epuration or use of catecholamines will also be recorded. In the 3-month and 12-month.

SUMMARY:
The purpose of this study is to assess the impact of Acute Kidney Injury (AKI) characteristics on long-term renal prognosis in Intensive Care Unit (ICU) patients.

DETAILED DESCRIPTION:
This study will be a multicentre prospective observational study. The MAKE evaluation after different kind of Acute Kidney Injury (MAKI) study will be conducted in 4 Intensive Care Units (ICU) in Clermont-Ferrand, France.

An information form about the study will be given to each ICU patients hospitalized more than 24 hours. This form will be given to their support person if it is not possible. Data during ICU stay related to renal function of patients included in the study will be collected. If available data related to their baseline kidney function (before ICU hospitalisation) will be collected.

The patients will be classified into 3 groups based on the occurrence of AKI and its duration: 1) patients without AKI during their stay, 2) patients who had a transient AKI episode (defined as recovery within 48 hours of onset), and 3) patients who had a persistent AKI episode during their stay.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are hospitalized for more than 24 hours in ICU will be eligible to participate in the study.

Exclusion Criteria:

* patients who are younger than 18 years,
* those who are pregnant,
* those who have chronic extrarenal epuration before their admission to the ICU,
* those who are admitted for kidney transplantation,
* those under the safeguard of justice, and those who refuse to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The MAKI study will recruit a large population of ICU patients. Patients who are hospitalized for more than 24 hours in ICU will be eligible to participate in the study. The MAKE evaluation after different kind of Acute Kidney Injury (MAKI) study will be conducted in 4 ICUs in Clermont-Ferrand, France. All ICU units include both medical and surgical patient recruitment.
  The patients will be classified into 3 groups based on the occurrence of AKI and its duration: 1) patients without AKI during their stay, 2) patients who had a transient AKI episode (defined as recovery within 48 hours of onset), and 3) patients who had a persistent AKI episode during their stay.
Sampling Method: Non-Probability Sample
Enrollment: 860 (Estimated)
Dates: Start 2022-11-22 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Kidney Event (MAKE) outcome at 3-month | 3 months after the onset of AKI or 3 months after ICU admission for patients without occurrence of AKI during their ICU stay.
  MAKE includes three main components:
  * Chronic Kidney Disease (CKD) occurrence or progression: Among patients who did not have CKD prior to the hospitalization, CKD occurrence is defined as a 25% or greater reduction in estimated GFR at 3-month or 12-month posthospitalization measurements compared to the baseline estimation and achievement of CKD stage 3 or higher. Progression of CKD in patients with pre-existing CKD at the time of hospitalization (preadmission estimated GFR < 60ml/min/1.73m2) is defined as a 50% or greater reduction in estimated GFR at 3-month or 12-month posthospitalization measurements and achievement of CKD stage 5 or receipt of chronic extrarenal epuration or kidney transplant (15,47).
  * Need for chronic extrarenal epuration
  * Death

SECONDARY OUTCOMES:
MAKE outcome at 12-month | 12 months after the onset of AKI or 12 months after ICU admission for patients without occurrence of AKI during their ICU stay.
  MAKE includes three main components:
  * Chronic Kidney Disease (CKD) occurrence or progression: Among patients who did not have CKD prior to the hospitalization, CKD occurrence is defined as a 25% or greater reduction in estimated GFR at 3-month or 12-month posthospitalization measurements compared to the baseline estimation and achievement of CKD stage 3 or higher. Progression of CKD in patients with pre-existing CKD at the time of hospitalization (preadmission estimated GFR < 60ml/min/1.73m2) is defined as a 50% or greater reduction in estimated GFR at 3-month or 12-month posthospitalization measurements and achievement of CKD stage 5 or receipt of chronic extrarenal epuration or kidney transplant.
  * Need for chronic extrarenal epuration
  * Death
CKD (occurence or progression if present before AKI) at 3-month | 3 months after the onset of AKI or 3 months after ICU admission for patients without occurrence of AKI during their ICU stay.
  Chronic Kidney Disease (CKD) occurrence or progression: Among patients who did not have CKD prior to the hospitalization, CKD occurrence is defined as a 25% or greater reduction in estimated GFR at 3-month or 12-month posthospitalization measurements compared to the baseline estimation and achievement of CKD stage 3 or higher. Progression of CKD in patients with pre-existing CKD at the time of hospitalization (preadmission estimated GFR < 60ml/min/1.73m2) is defined as a 50% or greater reduction in estimated GFR at 3-month or 12-month posthospitalization measurements and achievement of CKD stage 5 or receipt of chronic extrarenal epuration or kidney transplant.
CKD (occurence or progression if present before AKI) at 12-month | 12 months after the onset of AKI or 12 months after ICU admission for patients without occurrence of AKI during their ICU stay.
  Chronic Kidney Disease (CKD) occurrence or progression: Among patients who did not have CKD prior to the hospitalization, CKD occurrence is defined as a 25% or greater reduction in estimated GFR at 3-month or 12-month posthospitalization measurements compared to the baseline estimation and achievement of CKD stage 3 or higher. Progression of CKD in patients with pre-existing CKD at the time of hospitalization (preadmission estimated GFR < 60ml/min/1.73m2) is defined as a 50% or greater reduction in estimated GFR at 3-month or 12-month posthospitalization measurements and achievement of CKD stage 5 or receipt of chronic extrarenal epuration or kidney transplant.
chronic extra-renal epuration or kidney transplantation at 3-month | 3 months after the onset of AKI or 3 months after ICU admission for patients without occurrence of AKI during their ICU stay.
  This information will be recorded through a phone call.
chronic extra-renal epuration or kidney transplantation at 12-month | 12 months after the onset of AKI or 12 months after ICU admission for patients without occurrence of AKI during their ICU stay.
  This information will be recorded through a phone call.
Death occurence at 3-months | 3 months after the onset of AKI or 3 months after ICU admission for patients without occurrence of AKI during their ICU stay.
  This information will be recorded through a phone call.
Death occurence at 12-months | 12 months after the onset of AKI or 12 months after ICU admission for patients without occurrence of AKI during their ICU stay.
  This information will be recorded through a phone call.
MAKE outcome at 3-month according to the main pathophysiological mechanism of AKI: pre-renal, organic, or obstructive | 3 months after the AKI onset.
  The main pathophysiological mechanisms will be defined retrospectively by a board of nephrologist experts.
MAKE outcome at 12-month according to the main pathophysiological mechanism of AKI: pre-renal, organic, or obstructive | 12 months after the AKI onset.
  The main pathophysiological mechanisms will be defined retrospectively by a board of nephrologist experts.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Lautrette, Principal Investigator — University Hospital, Clermont-Ferrand; Cécile Gosset, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (2):
- France (2):
  - Centre Jean-Perrin, Clermont-Ferrand
  - CHU clermont-ferrand, Clermont-Ferrand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hoste EA, Bagshaw SM, Bellomo R, Cely CM, Colman R, Cruz DN, Edipidis K, Forni LG, Gomersall CD, Govil D, Honore PM, Joannes-Boyau O, Joannidis M, Korhonen AM, Lavrentieva A, Mehta RL, Palevsky P, Roessler E, Ronco C, Uchino S, Vazquez JA, Vidal Andrade E, Webb S, Kellum JA. Epidemiology of acute kidney injury in critically ill patients: the multinational AKI-EPI study. Intensive Care Med. 2015 Aug;41(8):1411-23. doi: 10.1007/s00134-015-3934-7. Epub 2015 Jul 11. PMID 26162677
- [Background] Lewington AJ, Cerda J, Mehta RL. Raising awareness of acute kidney injury: a global perspective of a silent killer. Kidney Int. 2013 Sep;84(3):457-67. doi: 10.1038/ki.2013.153. Epub 2013 May 1. PMID 23636171
- [Background] Chawla LS, Bellomo R, Bihorac A, Goldstein SL, Siew ED, Bagshaw SM, Bittleman D, Cruz D, Endre Z, Fitzgerald RL, Forni L, Kane-Gill SL, Hoste E, Koyner J, Liu KD, Macedo E, Mehta R, Murray P, Nadim M, Ostermann M, Palevsky PM, Pannu N, Rosner M, Wald R, Zarbock A, Ronco C, Kellum JA; Acute Disease Quality Initiative Workgroup 16.. Acute kidney disease and renal recovery: consensus report of the Acute Disease Quality Initiative (ADQI) 16 Workgroup. Nat Rev Nephrol. 2017 Apr;13(4):241-257. doi: 10.1038/nrneph.2017.2. Epub 2017 Feb 27. PMID 28239173
- [Background] Truche AS, Ragey SP, Souweine B, Bailly S, Zafrani L, Bouadma L, Clec'h C, Garrouste-Orgeas M, Lacave G, Schwebel C, Guebre-Egziabher F, Adrie C, Dumenil AS, Zaoui P, Argaud L, Jamali S, Goldran Toledano D, Marcotte G, Timsit JF, Darmon M. ICU survival and need of renal replacement therapy with respect to AKI duration in critically ill patients. Ann Intensive Care. 2018 Dec 17;8(1):127. doi: 10.1186/s13613-018-0467-6. PMID 30560526
- [Background] Khwaja A. KDIGO clinical practice guidelines for acute kidney injury. Nephron Clin Pract. 2012;120(4):c179-84. doi: 10.1159/000339789. Epub 2012 Aug 7. No abstract available. PMID 22890468
- [Background] Perinel S, Vincent F, Lautrette A, Dellamonica J, Mariat C, Zeni F, Cohen Y, Tardy B, Souweine B, Darmon M. Transient and Persistent Acute Kidney Injury and the Risk of Hospital Mortality in Critically Ill Patients: Results of a Multicenter Cohort Study. Crit Care Med. 2015 Aug;43(8):e269-75. doi: 10.1097/CCM.0000000000001077. PMID 25962084
- [Background] Coelho S, Fonseca JN, Gameiro J, Jorge S, Velosa J, Lopes JA. Transient and persistent acute kidney injury in acute liver failure. J Nephrol. 2019 Apr;32(2):289-296. doi: 10.1007/s40620-018-00568-w. Epub 2018 Dec 19. PMID 30569444
- [Background] Kim CS, Bae EH, Ma SK, Kweon SS, Kim SW. Impact of Transient and Persistent Acute Kidney Injury on Chronic Kidney Disease Progression and Mortality after Gastric Surgery for Gastric Cancer. PLoS One. 2016 Dec 9;11(12):e0168119. doi: 10.1371/journal.pone.0168119. eCollection 2016. PMID 27936153
- [Background] Bhatraju PK, Mukherjee P, Robinson-Cohen C, O'Keefe GE, Frank AJ, Christie JD, Meyer NJ, Liu KD, Matthay MA, Calfee CS, Christiani DC, Himmelfarb J, Wurfel MM. Acute kidney injury subphenotypes based on creatinine trajectory identifies patients at increased risk of death. Crit Care. 2016 Nov 17;20(1):372. doi: 10.1186/s13054-016-1546-4. PMID 27852290
- [Background] Horne KL, Packington R, Monaghan J, Reilly T, McIntyre CW, Selby NM. The effects of acute kidney injury on long-term renal function and proteinuria in a general hospitalised population. Nephron Clin Pract. 2014;128(1-2):192-200. doi: 10.1159/000368243. Epub 2014 Nov 28. PMID 25472765
- [Background] Horne KL, Packington R, Monaghan J, Reilly T, Selby NM. Three-year outcomes after acute kidney injury: results of a prospective parallel group cohort study. BMJ Open. 2017 Mar 29;7(3):e015316. doi: 10.1136/bmjopen-2016-015316. PMID 28360257
- [Background] Forni LG, Darmon M, Ostermann M, Oudemans-van Straaten HM, Pettila V, Prowle JR, Schetz M, Joannidis M. Renal recovery after acute kidney injury. Intensive Care Med. 2017 Jun;43(6):855-866. doi: 10.1007/s00134-017-4809-x. Epub 2017 May 2. PMID 28466146
- [Background] Heung M, Steffick DE, Zivin K, Gillespie BW, Banerjee T, Hsu CY, Powe NR, Pavkov ME, Williams DE, Saran R, Shahinian VB; Centers for Disease Control and Prevention CKD Surveillance Team. Acute Kidney Injury Recovery Pattern and Subsequent Risk of CKD: An Analysis of Veterans Health Administration Data. Am J Kidney Dis. 2016 May;67(5):742-52. doi: 10.1053/j.ajkd.2015.10.019. Epub 2015 Dec 12. PMID 26690912
- [Background] See EJ, Toussaint ND, Bailey M, Johnson DW, Polkinghorne KR, Robbins R, Bellomo R. Risk factors for major adverse kidney events in the first year after acute kidney injury. Clin Kidney J. 2019 Dec 20;14(2):556-563. doi: 10.1093/ckj/sfz169. eCollection 2021 Feb. PMID 33623679
- [Background] Bucaloiu ID, Kirchner HL, Norfolk ER, Hartle JE 2nd, Perkins RM. Increased risk of death and de novo chronic kidney disease following reversible acute kidney injury. Kidney Int. 2012 Mar;81(5):477-85. doi: 10.1038/ki.2011.405. Epub 2011 Dec 7. PMID 22157656
- [Background] Uchino S, Bellomo R, Bagshaw SM, Goldsmith D. Transient azotaemia is associated with a high risk of death in hospitalized patients. Nephrol Dial Transplant. 2010 Jun;25(6):1833-9. doi: 10.1093/ndt/gfp624. Epub 2010 Jan 6. PMID 20054022
- [Background] Pannu N, James M, Hemmelgarn B, Klarenbach S; Alberta Kidney Disease Network. Association between AKI, recovery of renal function, and long-term outcomes after hospital discharge. Clin J Am Soc Nephrol. 2013 Feb;8(2):194-202. doi: 10.2215/CJN.06480612. Epub 2012 Nov 2. PMID 23124779
- [Background] Sood MM, Shafer LA, Ho J, Reslerova M, Martinka G, Keenan S, Dial S, Wood G, Rigatto C, Kumar A; Cooperative Antimicrobial Therapy in Septic Shock (CATSS) Database Research Group. Early reversible acute kidney injury is associated with improved survival in septic shock. J Crit Care. 2014 Oct;29(5):711-7. doi: 10.1016/j.jcrc.2014.04.003. Epub 2014 Apr 18. PMID 24927984
- [Background] Uhel F, Peters-Sengers H, Falahi F, Scicluna BP, van Vught LA, Bonten MJ, Cremer OL, Schultz MJ, van der Poll T; MARS consortium. Mortality and host response aberrations associated with transient and persistent acute kidney injury in critically ill patients with sepsis: a prospective cohort study. Intensive Care Med. 2020 Aug;46(8):1576-1589. doi: 10.1007/s00134-020-06119-x. Epub 2020 Jun 8. PMID 32514599
- [Background] Schiffl H, Lang SM, Fischer R. Long-term outcomes of survivors of ICU acute kidney injury requiring renal replacement therapy: a 10-year prospective cohort study. Clin Kidney J. 2012 Aug;5(4):297-302. doi: 10.1093/ckj/sfs070. PMID 25874084
- [Background] Goldstein SL, Chawla L, Ronco C, Kellum JA. Renal recovery. Crit Care. 2014 Jan 6;18(1):301. doi: 10.1186/cc13180. PMID 24393370
- [Background] Chew STH, Hwang NC. Acute Kidney Injury After Cardiac Surgery: A Narrative Review of the Literature. J Cardiothorac Vasc Anesth. 2019 Apr;33(4):1122-1138. doi: 10.1053/j.jvca.2018.08.003. Epub 2018 Aug 7. PMID 30228051
- [Background] Kellum JA. Persistent Acute Kidney Injury. Crit Care Med. 2015 Aug;43(8):1785-6. doi: 10.1097/CCM.0000000000001102. No abstract available. PMID 26181122
- [Background] Ronco C, Bellomo R, Kellum JA. Acute kidney injury. Lancet. 2019 Nov 23;394(10212):1949-1964. doi: 10.1016/S0140-6736(19)32563-2. PMID 31777389
- [Background] Pickering JW, Frampton CM, Endre ZH. Evaluation of trial outcomes in acute kidney injury by creatinine modeling. Clin J Am Soc Nephrol. 2009 Nov;4(11):1705-15. doi: 10.2215/CJN.00820209. Epub 2009 Sep 3. PMID 19729431
- [Background] Pickering JW, Endre ZH. Baseline creatinine: where to from here? Nephrol Dial Transplant. 2011 Jun;26(6):2056; author reply 2056-7. doi: 10.1093/ndt/gfr099. Epub 2011 Mar 18. No abstract available. PMID 21421592
- [Background] Zavada J, Hoste E, Cartin-Ceba R, Calzavacca P, Gajic O, Clermont G, Bellomo R, Kellum JA; AKI6 investigators. A comparison of three methods to estimate baseline creatinine for RIFLE classification. Nephrol Dial Transplant. 2010 Dec;25(12):3911-8. doi: 10.1093/ndt/gfp766. Epub 2010 Jan 25. PMID 20100732
- [Background] De Rosa S, Samoni S, Ronco C. Creatinine-based definitions: from baseline creatinine to serum creatinine adjustment in intensive care. Crit Care. 2016 Mar 15;20:69. doi: 10.1186/s13054-016-1218-4. PMID 26983854
- [Background] Ichai C, Vinsonneau C, Souweine B, Armando F, Canet E, Clec'h C, Constantin JM, Darmon M, Duranteau J, Gaillot T, Garnier A, Jacob L, Joannes-Boyau O, Juillard L, Journois D, Lautrette A, Muller L, Legrand M, Lerolle N, Rimmele T, Rondeau E, Tamion F, Walrave Y, Velly L; Societe francaise d'anesthesie et de reanimation (Sfar); Societe de reanimation de langue francaise (SRLF); Groupe francophone de reanimation et urgences pediatriques (GFRUP); Societe francaise de nephrologie (SFN). Acute kidney injury in the perioperative period and in intensive care units (excluding renal replacement therapies). Ann Intensive Care. 2016 Dec;6(1):48. doi: 10.1186/s13613-016-0145-5. Epub 2016 May 27. PMID 27230984
- [Background] Bhatraju PK, Zelnick LR, Chinchilli VM, Moledina DG, Coca SG, Parikh CR, Garg AX, Hsu CY, Go AS, Liu KD, Ikizler TA, Siew ED, Kaufman JS, Kimmel PL, Himmelfarb J, Wurfel MM. Association Between Early Recovery of Kidney Function After Acute Kidney Injury and Long-term Clinical Outcomes. JAMA Netw Open. 2020 Apr 1;3(4):e202682. doi: 10.1001/jamanetworkopen.2020.2682. PMID 32282046
- [Background] Jones J, Holmen J, De Graauw J, Jovanovich A, Thornton S, Chonchol M. Association of complete recovery from acute kidney injury with incident CKD stage 3 and all-cause mortality. Am J Kidney Dis. 2012 Sep;60(3):402-8. doi: 10.1053/j.ajkd.2012.03.014. Epub 2012 Apr 27. PMID 22541737
- [Background] Ye N, Xu Y, Bellomo R, Gallagher M, Wang AY. Effect of nephrology follow-up on long-term outcomes in patients with acute kidney injury: A systematic review and meta-analysis. Nephrology (Carlton). 2020 Aug;25(8):607-615. doi: 10.1111/nep.13698. Epub 2020 Feb 18. PMID 32020718